CLINICAL TRIAL: NCT00080626
Title: A Pilot Study Assessing Patterns of Response or Resistance to Preoperative Dose Dense Docetaxel in Women With Newly Diagnosed Breast Cancer
Brief Title: Neoadjuvant Docetaxel in Treating Women With Newly Diagnosed Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0266; P50CA088843 (NIH); P30CA006973 (NIH); NA_00040559 (Other: JHM IRB); JHOC-03012301 (Other: SKCCC); JHOC-J0266 (Other: SKCCC); CDR0000346460 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pegfilgrastim; Docetaxel; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Docetaxel (Experimental): Neoadjuvant therapy with docetaxel (IV, 100 mg/m2, every 14 days with growth factor support with pegfilgrastim) for a total of 4 cycles prior to conventional surgery for breast cancer.
  Interventions: Biological: pegfilgrastim; Drug: docetaxel; Procedure: conventional surgery; Procedure: neoadjuvant therapy

INTERVENTIONS:
Biological: pegfilgrastim — 6 mg injection on day 1 of each cycle
  Other Names: Neulasta
Drug: docetaxel — 100 mg per meter-squared, every 14 days for 4 cycles
  Other Names: Taxotere
Procedure: conventional surgery — lumpectomy or mastectomy at end of treatment
  Other Names: definitive surgery
Procedure: neoadjuvant therapy — treatment prior to definitive breast surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving a chemotherapy drug before surgery may shrink the tumor so that it can be removed.

PURPOSE: This phase II trial is studying how well neoadjuvant docetaxel works in treating women who are undergoing surgery for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Correlate baseline and change in apoptosis and proliferation with clinical and pathological response to neoadjuvant docetaxel followed by surgery in women with newly diagnosed breast cancer.

Secondary

* Correlate baseline and change in fludeoxyglucose F 18 positron emission tomography uptake with clinical and pathological response in patients treated with this regimen.
* Correlate baseline and change in gene expression profiles with clinical and pathological response in patients treated with this regimen.
* Correlate baseline and change in tumor and serum proteomic patterns with clinical and pathological response in patients treated with this regimen.

OUTLINE: This is a pilot study.

* Neoadjuvant chemotherapy: Patients receive docetaxel IV over 1 hour on day 1 and pegfilgrastim subcutaneously (SC) on day 2. Treatment repeats every 14 days for 4 courses in the absence of disease progression or unacceptable toxicity.
* Surgery: Within 2-4 weeks after the completion of 4 courses of docetaxel, patients undergo breast-conserving surgery or a mastectomy at the discretion of the treating surgeon. Patients may receive additional chemotherapy prior to surgery at the discretion of the treating physician.
* Adjuvant chemotherapy: Patients receive adjuvant chemotherapy at the discretion of the treating physician.
* Radiotherapy: Patients undergo radiotherapy after the completion of all chemotherapy at the discretion of the treating physician.
* Hormonal therapy: Patients with estrogen- and/or progesterone-positive tumors receive hormonal therapy after the completion of chemotherapy and all local therapies at the discretion of the treating physician.

Patients are followed every 6 months.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed infiltrating carcinoma of the breast

  * Unresected clinical stage T1c, T2, T3, or T4 lesion, any N
* Newly diagnosed disease

  * Diagnostic mammogram and an ultrasound of the affected breast within 3 months before study entry
  * Mammogram of the contralateral breast within 6 months before study entry
* Clinically measurable disease
* Hormone receptor status:

  * Immunohistochemical staining for estrogen and progesterone and HER2/neu receptors must be obtained on initial diagnostic material

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 8 g/dL

Hepatic

* Bilirubin no greater than 1.5 times normal

Renal

* Creatinine no greater than 1.5 times normal

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No medical condition that would put the patient at unnecessary risk of potentially serious complications during study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for current breast cancer

Endocrine therapy

* At least 1 month since prior tamoxifen or raloxifene for breast cancer prevention
* No prior endocrine therapy for current breast cancer

Radiotherapy

* No prior radiotherapy for current breast cancer

Surgery

* Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2003-08-11 (Actual); Primary Completion 2006-05-01 (Actual); Study Completion 2006-05-01 (Actual)

PRIMARY OUTCOMES:
Correlation between change in apoptosis and proliferation with response after definitive surgery | Definitive surgery

SECONDARY OUTCOMES:
Correlation between change in fludeoxyglucose F 18 positron emission tomography uptake with response after definitive surgery | Definitive surgery

CONTACTS AND LOCATIONS:
Overall Officials: Vered Stearns, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States